CLINICAL TRIAL: NCT01132326
Title: A Multi-center, Open-label Study to Assess the Long-term Safety of Droxidopa in Subjects With Primary Autonomic Failure, Dopamine Beta Hydroxylase Deficiency or Non-Diabetic Neuropathy and Symptomatic Neurogenic Orthostatic Hypotension
Brief Title: Clinical Study of Droxidopa in Patients With Neurogenic Orthostatic Hypotension (NOH) (Droxi-304)
Acronym: NOH304
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Droxidopa NOH304
Record Dates: First submitted 2009-09-09; First posted 2010-05-28 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Primary Autonomic Failure; Dopamine Beta Hydroxylase Deficiency; Non-Diabetic Neuropathy; Neurogenic Orthostatic Hypotension
Keywords: Symptomatic NOH
MeSH Terms: conditions — dopamine beta hydroxylase deficiency | interventions — Droxidopa; 3,4-dihydroxyphenylserine aldolase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Droxidopa (Experimental): Open-Label Droxidopa
  Interventions: Drug: Droxidopa

INTERVENTIONS:
Drug: Droxidopa — Oral, 100, 200, 300, 400, 500, 600 mg TID, 12 months
  Other Names: L-threo-3,4-dihydroxyphenylserine; L-threo-DOPS

SUMMARY:
Symptomatic NOH in patients with primary autonomic failure is thought to be a consequence of norepinephrine depletion leading to a diminished capacity to effect an appropriate cardiovascular response to an orthostatic challenge resulting in symptomatic cerebral-hypoperfusion. Droxidopa augments norepinephrine levels which should lead to improved cerebral perfusion following orthostatic challenge thereby reducing the symptoms of NOH. The present study will evaluate the long-term safety of droxidopa.

DETAILED DESCRIPTION:
This is a Phase III, multi-center, open-label study designed to evaluate the long-term safety of droxidopa in subjects with neurogenic orthostatic hypotension (NOH) associated with Primary Autonomic Failure, Dopamine Beta Hydroxylase Deficiency or Non-Diabetic Autonomic Neuropathy.

Patients will be initially treated with droxidopa at their individualized dose identified during the titration phase in Protocol 301. Patients will not require adjustment of their dose, unless their physician feels a dose change will benefit their symptoms, or side effects. At any point in the study a patient's physician may elect to titrate the subject to a higher or lower dose if they feel additional benefit can be safely derived or to deal with any unwanted side-effect.

Patients will return to the clinic for study visits at 1, 3, 6, 9 and 12 months (± 1 week allowed for 1 month visit, ± 2 weeks allowed for subsequent study visits). Patients who prematurely withdraw from the study will be asked to attend the study center for a final assessment At the conclusion of the 12 month treatment period, all patients who benefit from treatment with droxidopa will be offered the option to continue to receive open-label droxidopa through a separate access program.

At any time during the study, patients can schedule a visit with their study physician if they experience a worsening of symptoms and wish to have their dose adjusted or to remove themselves from the trial.

Patients who decide to terminate their participation in the study will receive a phone call 1 month after leaving the trial to follow-up on any new or ongoing adverse events (AEs).

It is a recognized best practice that patients with neurogenic orthostatic hypotension are advised not to lay fully supine because of the associated increased risk of supine hypertension inherent with their condition. Patients participating in this study should be advised to sleep in a semi-recumbent position. .

Patients will attend the study center as out-patients. Patients will be identified using the unique identification number assigned during Protocol 301.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, each patient must fulfill the following criteria:

* Demonstrated a symptomatic response (an improvement of at least 1 point in Item #1 of the OHSA) to treatment with droxidopa during open-label titration in Droxidopa Protocol 301 ;
* Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care.

Exclusion Criteria:

Patients are not eligible for this study if they fulfill one or more of the following criteria:

* Currently taking vasoconstricting agents such as ephedrine, dihydroergotamine, or midodrine; patients taking vasoconstricting agents such as ephedrine, dihydroergotamine, or midodrine must stop taking these drugs at least 2 days or 5 half-lives (whichever is longer) prior to their study entry visit (Visit 1).
* Currently taking anti-hypertensive medication; the use of short-acting anti-hypertensive medications at bedtime is permitted.
* Currently taking tri-cyclic antidepressant medication or other norepinephrine re-uptake inhibitors;
* Have changed dose, frequency and or type of prescribed medication, within two weeks of starting droxidopa treatment within Protocol 304, with the following exceptions:

  * vasoconstricting agents such as ephedrine, dihydroergotamine, or midodrine (see exclusion a),
  * short courses of antibiotics or other medications/treatments that do not interfere with, or exacerbate the patient's condition under study.
* History of known or suspected drug or substance abuse;
* Women of childbearing potential who are not using a medically accepted contraception;

  * Reproductive potential: Female subjects should be either post-menopausal (amenorrhoea for at least 12 consecutive months), surgically sterile, or women of child-bearing potential (WOCP) who are using or agree to use acceptable methods of contraception. Acceptable contraceptives include intrauterine devices (IUDs), hormonal contraceptives (oral, depot, patch or injectable) and double barrier methods such as condoms or diaphragms with spermicidal gel or foam.
  * For WOCP a serum beta HCG pregnancy test must be conducted at screening, and a urine pregnancy test must be conducted at baseline and study termination; the results must be negative at screening and at baseline for the patient to receive study medication. WOCP must be advised to use acceptable contraceptives throughout the study period and for 30 days after the last dose of investigational product. If hormonal contraceptives are used they should be taken according to the package insert. WOCP who are not currently sexually active must agree to use acceptable contraception, as defined above, if they decide to become sexually active during the period of the study and for 30 days after the last dose of investigational product.
* Sexually active males whose partner is a WOCP and who do not agree to use condoms for the duration of the study and for 30 days after the last dose;
* Women who are pregnant or breast feeding;
* Known or suspected hypersensitivity to the study medication or any of its ingredients;
* Pre-existing, sustained, severe hypertension (BP greater than or equal to 180/110 mmHg in the sitting position);
* Have atrial fibrillation or, in the investigator's opinion, have any other significant cardiac arrhythmia;
* Any other significant systemic, hepatic, cardiac or renal illness;
* Diabetes mellitus or insipidus;
* Have a history of closed angle glaucoma;
* Have a known or suspected malignancy;
* Patients with known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug;
* In the investigator's opinion, have clinically significant abnormalities on clinical examination or laboratory testing;
* In the investigator's opinion, are unable to adequately co-operate because of individual or family situation;
* In the investigator's opinion, are suffering from a mental disorder that interferes with the diagnosis and/or with the conduct of the study, e.g. schizophrenia, major depression, dementia;
* Are not able or willing to comply with the study requirements for the duration of the study;
* Have participated in another clinical trial with an investigational agent other than droxidopa (including named patient or compassionate use protocol) within 4 weeks before starting droxidopa treatment within Protocol 304;
* Previous enrolment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2009-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, MD, Principal Investigator — NYU Langone Health

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Droxidopa
Started | 350
Completed | 132
Not Completed | 218
Not completed — Lack of Efficacy | 25
Not completed — Adverse Event | 37
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 16
Not completed — Withdrawal by Subject | 40
Not completed — Physician Decision | 10
Not completed — Study Termination | 80
Not completed — Declining Health | 1
Not completed — Pregnancy | 1
Not completed — Caregiver Withdrew Consent | 1
Not completed — Death | 5
Not completed — Subject Unable to Come To Visits | 1

BASELINE CHARACTERISTICS:
Arm/Group | Droxidopa
Number analyzed (Participants) | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (15.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 214
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 344
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 263
  Europe | 87
Primary Clinical Diagnosis [Number; unit: participants]
  Parkinson's Disease | 232
  Multiple System Atrophy | 33
  Pure Autonomic Failure | 68
  Dopamine Beta-Hydroxylase Deficiency | 0
  Non-Diabetic Autonomic Neuropathy | 8
  Other | 7
  Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Patients With Treatment-emergent Adverse Events
Description: Number of patients reporting any treatment emergent adverse events (SAE and or AEs) during the study
Time Frame: up to 2 years
Measure: Number; unit: participants
Arm/Group | Droxidopa
Number analyzed (Participants) | 350
participants | 263

ADVERSE EVENTS:
Arm/Group | Droxidopa
Serious Adverse Events (participants affected / at risk) | 83/350
Other Adverse Events (participants affected / at risk) | 178/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa (N=350)
Syncope (Nervous system disorders) | 10 (11)
Transient ischaemic attack (Nervous system disorders) | 3 (3)
Cerebral infarct (Nervous system disorders) | 2 (2)
Multiple system atrophy (Nervous system disorders) | 2 (2)
Parkinson's disease (Nervous system disorders) | 2 (2)
Altered state of conciousness (Nervous system disorders) | 1 (1)
Brain edema (Nervous system disorders) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Presyncopy (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 7 (10)
Sepsis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Localized infection (Infections and infestations) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Peridiverticular abscess (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 3 (5)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 2 (2)
Aortic aneurysm (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hemorrhagic infarction (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1)
Respiratory failure- (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Supra-ventricular tachycardia (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Hypovolemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 2 (2)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Hyperthermia (General disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 2 (2)
Suicide attempt (Psychiatric disorders) | 2 (2)
Acute psychosis (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Psychiatric disorder (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Colitis ischemia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Inter-vertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parathyroid tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa (N=350)
Headache (Nervous system disorders) | 42 (59)
Syncope (Nervous system disorders) | 35 (44)
Dizziness (Nervous system disorders) | 34 (54)
Fall (Injury, poisoning and procedural complications) | 80 (157)
Contusion (Injury, poisoning and procedural complications) | 18 (40)
Urinary tract infection (Infections and infestations) | 45 (107)
Nausea (Gastrointestinal disorders) | 23 (27)
Fatigue (General disorders) | 28 (30)
Asthenia (General disorders) | 20 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less